CLINICAL TRIAL: NCT07185945
Title: Phase II Trial of Zanzalintinib for Advanced Urothelial Carcinoma Progressing After Prior Therapy
Brief Title: Zanzalintinib for Advanced Urothelial Carcinoma Progressing After Prior Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guru Sonpavde (Other)
Collaborators: Exelixis (Industry); Advent Health (Unknown)
Responsible Party: Sponsor-Investigator, Guru Sonpavde, sponsor-investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU23-633
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Urothelial Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanzalintinib (Experimental): All subjects will receive Zanzalintinib 60 mg orally once daily until progression per RECIST 1.1 or intolerable toxicities or patient/investigator decision to discontinue study therapy.
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — 60 mg orally once daily

SUMMARY:
This is a Phase II, single arm study. All subjects will receive Zanzalintinib 60 mg orally once daily until progression per RECIST 1.1 or intolerable toxicities or patient/investigator decision to discontinue study therapy. Radiology imaging will be performed every 8 weeks for 3 timepoints then every 12 weeks thereafter. A window of ± 7 days may be applied to all study visits to accommodate observed holidays, inclement weather, scheduling conflicts etc.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 within 28 days prior to registration.
4. Histologically confirmed predominant urothelial carcinoma (T4b, N0, M0; any T, N1-N3, M0; any T, any N, M1). American Joint Committee on Cancer (AJCC) v8 staging manual. NOTE: must be locally advanced unresectable or metastatic.
5. Measurable disease according to RECIST 1.1 within 28 days prior to registration.
6. Progressive disease by RECIST 1.1 following 1 to 3 lines of prior therapy. NOTE: prior lines of therapy must include Enfortumab Vedotin (EV) [unless ineligible for EV] and PD(L)1 inhibitor [unless ineligible for PD(L)1 inhibitor]. Prior platinum-based chemotherapy and other agents are allowed but not required.
7. Prior cancer treatment must be completed ≥ 28 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen to Grade ≤ 1 or baseline. NOTE: Alopecia and sensory neuropathy of Grade ≤ 2 are acceptable.
8. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 14 days prior to registration.

   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   * Platelets (Plt) ≥ 100,000/mm3 (without transfusion within 14 days of screening laboratory sample collection)
   * Hemoglobin (Hgb) ≥ 8 g/dL (without transfusion within 14 days of screening laboratory sample collection)
   * Calculated creatinine clearance1 ≥ 40 mL/min
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3.0 × ULN for patients with Gilbert's disease
   * Aspartate aminotransferase (AST) ≤ 3 × ULN or ≤ 5 x ULN with liver metastases
   * Alanine aminotransferase (ALT) ≤ 3 × ULN or ≤ 5 x ULN with liver metastases
   * Alkaline Phosphatase (ALP) < 3 x ULN. NOTE: for patients with bone metastases ALP < 5x ULN
   * International Normalized Ratio (INR) or Prothrombin Time (PT)
   * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN
   * Urine protein to creatinine ratio (UPCR) ≤ 2 mg/mg (≤ 226.4 mg/mmol) creatinine
9. Females of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to registration. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from penile-vaginal intercourse or must use an effective method(s) of contraception. Males able to father a child who are sexually active with a female of childbearing potential must be willing to abstain from penile-vaginal intercourse or use an effective method(s) of contraception.
11. Subjects with known HIV-infection or acquired immunodeficiency syndrome (AIDS)-related illness on stable anti-retroviral therapy with a CD4+ T cell count ≥ 200/µL and undetectable viral load are eligible for this trial. NOTE: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to registration. Anti-retroviral therapies (ART) must have been received for at least 28 days prior to registration.
12. Subjects with a known chronic hepatitis B virus (HBV) infection, must have an undetectable HBV viral load on suppressive therapy, if indicated. Subjects with a history of hepatitis C virus (HCV) infection must have been treated and cured. For subjects with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial.
13. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. More than 3 lines of prior therapy (prior cisplatin-based perioperative chemotherapy within 1 year prior to subsequent therapy or registration, whichever comes first) and/or prior perioperative PD1 inhibitor within 12 weeks prior to subsequent therapy (or registration, whichever comes first) is considered a line of therapy).
2. Prior receipt of a VEGF inhibitor.
3. Prior receipt of zanzalintinib.
4. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 28 days before registration.
5. Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational therapy) within 28 days prior to Cycle 1 Day 1.
6. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors ) and platelet inhibitors (eg, clopidogrel) are allowed only if:

   * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 7 days before registration without clinically significant hemorrhagic complications from the anticoagulation regimen.

   NOTE: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to registration, whichever is longer.
7. Administration of a live, attenuated vaccine within 30 days before Cycle 1 Day 1.
8. Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 14 days before registration.
9. Pharmacologically uncompensated, symptomatic hypothyroidism
10. Current symptomatic central nervous system (CNS) metastases. NOTE: Patients with previously diagnosed CNS metastases are eligible if they have completed treatment and recovered from the acute effects of radiation therapy or surgery prior to registration, have tapered corticosteroid treatment to 10 mg/day or less and are neurologically stable.
11. Deep vein thrombosis or pulmonary embolism or prior clinically significant venous events per investigator discretion within 12 weeks prior to registration. NOTE: Subjects with a diagnosis of deep vein thrombosis (DVT) beyond 1 month earlier are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 7 days prior to registration without clinically significant hemorrhagic complications from the anticoagulation regimen. Subjects with a diagnosis of DVT within 24 weeks are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 7 days prior to registration without clinically significant hemorrhagic complications from the anticoagulation regimen.
12. Unstable or deteriorating cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension, defined as Systolic Blood Pressure > 140 mm Hg or Diastolic Blood Pressure > 90 mm Hg).
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 24 weeks before registration.
13. Left ventricular ejection fraction (LVEF) < 50% by Echocardiogram or Multigated Acquisition Scan (MUGA). NOTE: Results from an Echocardiogram or MUGA obtained within 1 year prior to registration may be used for eligibility.
14. Corrected QTcF by Frederica formula > 480 ms within 14 days of registration.
15. Prior history of myocarditis.
16. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI-tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 24 weeks prior to registration unless the cause of obstruction is definitively managed and subject is asymptomatic
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 24 weeks before registration. NOTE: Complete healing of an intra-abdominal abscess must be confirmed before Cycle 1 Day 1.
    * Known gastric or esophageal varices.
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 28 days prior to registration.
17. Clinically significant hematuria, hematemesis, or hemoptysis of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before registration.
18. Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
19. Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. NOTE: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following sponsor-investigator approval.
20. Active infection requiring systemic therapy. NOTE: Subjects receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
21. Inability to swallow tablets or ingest a suspension orally or by nasogastric (NG) or gastrostomy (PEG) tube.
22. Malabsorption syndrome.
23. Moderate to severe hepatic impairment (Child-Pugh B or C).
24. Major surgery within 8 weeks or minor surgery within 5 days before Cycle 1 Day 1. NOTE: Complete wound healing from major and minor surgery based on investigator discretion must have occurred prior to Cycle 1 Day 1.
25. Major radiation therapy < 14 days prior to Cycle 1 Day 1. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed < 14 days prior to registration.
26. Serious non-healing wound/ulcer/bone fracture. NOTE: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
27. Diagnosis of any other malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of trial therapy.
28. Requirement for hemodialysis or peritoneal dialysis.
29. History of solid organ or allogeneic stem cell transplant.
30. Pregnant or breastfeeding. NOTE: breast milk cannot be stored for future use while the subject is being treated on study.
31. History of severe allergic anaphylactic reactions to study drug or any of its' excipients.
32. History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  PFS is defined as the time from the date of study registration to the date of progression per RECIST 1.1 or death due to any cause, whichever occurs first.
Duration of Response (DOR) | 24 months
  DOR is defined as the time from the first documented response (PR or CR) until the time of progression per RECIST 1.1 or death due to any cause.
Overall survival (OS) | 24 months
  OS is defined as the time from the date of study registration to date of death due to any cause.
Number of Participants with Adverse Events | 24 months
  Adverse events will be assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — Advent Health Orlando